CLINICAL TRIAL: NCT04880733
Title: Acupuncture in the Emergency Department for Pain Management: A BraveNet Multi-Center Feasibility Study
Brief Title: Acupuncture in the Emergency Department for Pain Management
Acronym: ACUITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Vanderbilt University Medical Center (Other); University of California, San Diego (Other); Albert Einstein College of Medicine (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Jeffery Dusek, PhD, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: R01AT010598-01A1 (NIH)
Record Dates: First submitted 2021-04-30; First posted 2021-05-11 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Acupuncture; Pain Management; Emergency Department; Acute Pain
MeSH Terms: conditions — Agnosia; Emergencies; Acute Pain | interventions — Acupuncture Therapy; Pain Management

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data collector will be masked to study outcomes via electronic data collection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): This arm will receive acupuncture for pain management, and any pain medications will be delayed until after receipt of acupuncture.
  Interventions: Procedure: Acupuncture for pain management; Other: Usual care for pain management
- Usual Care (Active Comparator): This arm will receive usual care for pain management.
  Interventions: Other: Usual care for pain management

INTERVENTIONS:
Procedure: Acupuncture for pain management — A manualized acupuncture protocol will be performed by a licensed acupuncturist in the patient's emergency department room.
  Arms: Acupuncture
Other: Usual care for pain management — Patient will receive usual care for pain management.

SUMMARY:
Our goal is to use the R01 mechanism to conduct a two-arm multisite, feasibility RCT (Acupuncture vs Usual Care) to refine procedures for conducting a future fully powered multi-site RCT. The effort will be led by the BraveNet Coordinating Center at Einstein and include 3 BraveNet PBRN sites University Hospitals/ Case Western Reserve University (UH/Case), Vanderbilt University Medical Center (VUMC), and University of California-San Diego (UCSD). During Year 1 (Aim 1), we will develop the manualized acupuncture intervention with consensus from experts in the delivery of acupuncture for acute pain. At the end of Year 1 (prior to the start of the RCT), a study investigator meeting will be held to ensure consistent training of all study coordinators and acupuncturists to the study data collection, human subjects, intervention delivery, and reporting requirements. In Year 2-3 (Aim 2), we will enroll 165 participants (55 per site) into the randomized trial (1:1 assignment to Acupuncture or Usual Care) over a ~9-month enrollment period for each site. Sites will participate in the study sequentially, thus general findings from the implementation evaluation may be used to improve implementation at subsequent sites. Treatment outcomes include pain intensity, state anxiety and pain medication utilization within the ED (via EHR data extraction). In Aim 2a, 75 structured qualitative interviews of ED providers, staff, study acupuncturists (~10 per site) and acupuncture patients (~15 per site) and direct observation at each site will be used to identify barriers and facilitators of successful implementation. The Implementation Evaluation includes two broad categories of data: implementation outcomes (collected in Aim 2 as the feasibility study is conducted at each site) and explanatory factors (Aim 2a).

DETAILED DESCRIPTION:
The goal is to use the R01 mechanism to conduct a two-arm multisite, feasibility RCT (Acupuncture vs Usual Care) to refine procedures for conducting a future fully powered multi-site RCT. The effort will include the BraveNet Coordinating Center at Einstein and include 3 BraveNet PBRN sites University Hospitals/ Case Western Reserve University (UH/Case), Vanderbilt University Medical Center (VUMC), and University of California-San Diego (UCSD). During Year 1 (Aim 1), the investigators will develop the manualized acupuncture intervention with consensus from experts in the delivery of acupuncture for acute pain. Prior to the start of the RCT at all sites, study investigator meetings will be held to ensure consistent training of all study coordinators and acupuncturists to the study data collection, human subjects, intervention delivery, and reporting requirements. In Year 2-3 (Aim 2), the investigators will enroll 165 participants (55 per site) into the randomized trial (1:1 assignment to Acupuncture or Usual Care) over a ~9-month enrollment period for each site. Sites will participate in the study sequentially, thus general findings from the implementation evaluation may be used to improve implementation at subsequent sites. Study outcomes include responsive manualization of acupuncture intervention, recruitment, retention, patient adoption, patient acceptability, and provider acceptability. Measures will be collected including pain intensity, state anxiety and pain medication utilization within the ED (via EHR data extraction). In Aim 2a, 75 structured qualitative interviews of ED providers, staff, study acupuncturists (~10 per site) and acupuncture patients (~15 per site) and direct observation at each site will be used to identify barriers and facilitators of successful implementation. The Implementation Evaluation includes two broad categories of data: implementation outcomes (collected in Aim 2 as the feasibility study is conducted at each site) and explanatory factors (Aim 2a).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age
* Ability to communicate in English.
* Level 3, 4, 5 on triage rate scale
* Presentation with acute non-emergent (musculoskeletal, back, pelvic, non-cardiac chest, abdominal, flank or head) pain ≥4 on a 0-10-point NRS due to non-penetrating injury.

Exclusion Criteria:

* Fever exceeding 100° F
* Presenting with a chief complaint of a psychological / psychiatric concern
* Presenting with chief complaint of Migraine
* Patient arriving via ambulance or skipping triage
* Current Pregnancy
* Self-reported opioid medication taken orally within 4 hours
* Presenting with chief complaint of Joint Dislocation
* Presenting with chief complaint of Bone Fracture
* Confirmed or suspected COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-09-24 (Actual); Study Completion 2025-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery A Dusek, PhD, Principal Investigator — University California-Irvine; M. Diane McKee, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (4):
- United States (4):
  - University of California San Diego, La Jolla, California
  - Einstein School of Medicine, The Bronx, New York
  - University Hospitals/Case Western Reserve University- Cleveland Medical Center, Cleveland, Ohio
  - Vandebilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dusek JA, Kallenberg GA, Storrow AB, Hughes RM, Coyne CJ, Vago DR, Nielsen A, Karasz A, Kim RS, Surdam J, Segall T, Faryar KA, Dyer NL, Barton BA, McKee MD. Acupuncture in the emergency department (ACUITY): Results from a BraveNet multi-center feasibility randomized controlled trial. Integr Med Res. 2024 Dec;13(4):101095. doi: 10.1016/j.imr.2024.101095. Epub 2024 Oct 21. PMID 39640074
- [Derived] Nielsen A, Dyer NL, Lechuga C, McKee MD, Dusek JA. Fidelity to the acupuncture intervention protocol in the ACUpuncture In The EmergencY department for pain management (ACUITY) trial: Expanding the gold standard of STRICTA and CONSORT guidelines. Integr Med Res. 2024 Jun;13(2):101048. doi: 10.1016/j.imr.2024.101048. Epub 2024 May 10. PMID 38841077
- [Derived] Dusek JA, Kallenberg GA, Hughes RM, Storrow AB, Coyne CJ, Vago DR, Nielsen A, Karasz A, Kim RS, Surdam J, Segall T, McKee MD. Acupuncture in the emergency department for pain management: A BraveNet multi-center feasibility study. Medicine (Baltimore). 2022 Mar 4;101(9):e28961. doi: 10.1097/MD.0000000000028961. PMID 35244059
- [Derived] Nielsen A, Olson J, Quesada M, Zhu C, Raskin E, Vang B, Painovich J, Scott M, Xiong VJ, Dusek JA. Acupuncture intervention for acute pain in the Emergency Department trial: a consensus process. Acupunct Med. 2022 Aug;40(4):339-346. doi: 10.1177/09645284221076507. Epub 2022 Mar 1. PMID 35229658
- [Derived] Dyer NL, Surdam J, Dusek JA. A Systematic Review of Practiced-Based Research of Complementary and Integrative Health Therapies as Provided for Pain Management in Clinical Settings: Recommendations for the Future and a Call to Action. Pain Med. 2022 Jan 3;23(1):189-210. doi: 10.1093/pm/pnab151. PMID 34009391

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: May 3, 2021 - September 24, 2022 from three Emergency Departments
Pre-assignment Details: At the moment of consent,165 patients were randomized to group. However, 14 (7 per group) did not provide outcomes as detailed below. Complete participants were 151 at Post-Treatment.
  A sample of ED providers at the sites answered 2 questions on the appropriateness and helpfulness of acupuncture being provided in the Emergency Department.
  Individuals with direct exposure to ACUITY answered 2 more questions on satisfaction and burden of conducting ACUITY in their ED.
Groups:
- ED Staff/Providers: These were ED staff or providers who answered questions after their site had finished study recruitment.
Period: Participants in the RCT (Overall Study)
Arm/Group | Acupuncture | Usual Care | ED Staff/Providers
Started | 83 | 82 | 0
Received Acupuncture | 79 | 0 | 0
Received Usual Care | 0 | 82 | 0
Completed | 76 | 75 | 0
Not Completed | 7 | 7 | 0
Not completed — Data collection issue | 3 | 5 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0
Not completed — Delay due to ED imaging | 1 | 0 | 0
Not completed — Early discharge | 0 | 1 | 0
Period: ED Staff/Providers 6 Month Assessment
Arm/Group | Acupuncture | Usual Care | ED Staff/Providers
Started | 0 | 0 | 125
Completed Question 1 | 0 | 0 | 125
Completed Question 2 | 0 | 0 | 124
Completed Question 3 | 0 | 0 | 32
Completed Question 4 | 0 | 0 | 32
Completed | 0 | 0 | 124
Not Completed | 0 | 0 | 1
Not completed — Skipped question 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demographics and initial conditions of participants providing pre and post pain scores in part of the RCT.
  Or the demographics of the ED Staff/Providers who answered several questions at the 6 month point after recruitment in their ED was complete.
Groups:
- ED Staff/Providers: ED Staff and Providers were asked complete 2 questions about their perceptions of acupuncture in the ED.
  If the ED staff or providers had direct contact with the ACUITY study in their ED, then they were asked to complete 2 additional questions inquiring about how ACUITY may have impacted the ED.
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Usual Care | ED Staff/Providers | Total
Number analyzed (Participants) | 76 | 75 | 125 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (16.9) | 43.9 (17.4) | 37.6 (9.35) | 44.4 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 47 | 65 | 151
  Male | 37 | 28 | 60 | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity data not collected for the ED Staff/Providers Arm
  Participants
    number analyzed (Participants) | 76 | 75 | 0 | 151
    Hispanic or Latino | 9 | 11 | 0 | 20
    Not Hispanic or Latino | 67 | 64 | 0 | 131
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: individuals] — Population: Race/Ethnicity, Customized data not collected for the ED Staff/Providers Arm
  individuals
    White: number analyzed (Participants) | 76 | 75 | 0 | 151
    White | 37 | 28 |  | 65
    Black/AA: number analyzed (Participants) | 76 | 75 | 0 | 151
    Black/AA | 34 | 33 |  | 67
    Other: number analyzed (Participants) | 76 | 75 | 0 | 151
    Other | 5 | 14 |  | 19
Education [Count of Participants; unit: Participants] — Population: Education data not collected for the ED Staff/Providers Arm
  Participants
    number analyzed (Participants) | 76 | 75 | 0 | 151
    No high school diploma | 1 | 4 |  | 5
    High school or equivalent | 26 | 23 |  | 49
    Some college | 26 | 28 |  | 54
    College degree | 17 | 17 |  | 34
    Graduate or professional degree | 5 | 3 |  | 8
    Decline to answer | 1 | 0 |  | 1
Income [Count of Participants; unit: Participants] — Population: Income data not collected for the ED Staff/Providers Arm
  Participants
    number analyzed (Participants) | 76 | 75 | 0 | 151
    Less than $20,000 | 22 | 27 |  | 49
    $20,000 - $50,000 | 21 | 23 |  | 44
    $50,001 to $100,000 | 9 | 6 |  | 15
    $100,001 to $150,000 | 4 | 4 |  | 8
    More than $150,000 | 3 | 4 |  | 7
    Decline to answer | 17 | 11 |  | 28
Insurance [Count of Participants; unit: Participants] — Population: Insurance data not collected for the ED Staff/Providers Arm
  Participants
    number analyzed (Participants) | 76 | 75 | 0 | 151
    Medicare | 25 | 19 |  | 44
    Medicaid | 16 | 23 |  | 39
    Private insurance | 32 | 23 |  | 55
    No insurance | 2 | 6 |  | 8
    Decline to answer | 1 | 4 |  | 5
Location of Pain [Count of Participants; unit: Participants] — Population: Location of Pain data not collected for the ED Staff/Providers Arm
  Participants
    number analyzed (Participants) | 76 | 75 | 0 | 151
    Abdomen | 14 | 14 |  | 28
    Head | 7 | 6 |  | 13
    Flank | 3 | 2 |  | 5
    Chest | 2 | 2 |  | 4
    Back | 25 | 27 |  | 52
    Extremity | 16 | 22 |  | 38
    Neck | 1 | 0 |  | 1
    Multiple | 6 | 1 |  | 7
    Other | 2 | 1 |  | 3
Prior Acupuncture [Count of Participants; unit: Participants] — Population: Prior Acupuncture data not collected for the ED Staff/Providers Arm
  Participants
    number analyzed (Participants) | 76 | 75 | 0 | 151
    (all) | 19 | 17 |  | 36
Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — 0-10 Numeric Rating Scale of Pain Intensity (where "0" is No pain and "10" is maximal Pain) Population: Pain Intensity data not collected for the ED Staff/Providers Arm
  units on a scale
    number analyzed (Participants) | 76 | 75 | 0 | 151
    (all) | 7.4 (2.2) | 7.1 (2.3) |  | 7.3 (2.2)
Anxiety- acute [Mean (Standard Deviation); unit: units on a scale] — 0-10 Numeric Rating Scale of acute anxiety (where "0" is No anxiety and "10" is maximal anxiety) Population: Anxiety- acute data not collected for the ED Staff/Providers Arm
  units on a scale
    number analyzed (Participants) | 76 | 75 | 0 | 151
    (all) | 4.5 (3.4) | 4.1 (3.4) |  | 4.3 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Successful Recruitment of Participants Into the Study.
Description: The recruitment rate (# enrolled / # approached) were assessed for the overall study. Separate recruitment rates were calculated by site.
Time Frame: At Enrollment
Population: Patients who were eligible AND approached.
Measure: Number; unit: Percentage of participants enrolled
Groups:
- Total Approached: Total approached across all 3 sites
- University Hospitals/Case Western: Patients approached at University Hospitals/Case Western
- VUMC: Patients approached at VUMC
- UCSD: Patients approached at UCSD
Arm/Group | Total Approached | University Hospitals/Case Western | VUMC | UCSD
Number analyzed (Participants) | 632 | 220 | 300 | 112
Percentage of participants enrolled | 26.1 | 27.7 | 16.3 | 49.1

2. Secondary Outcome: Percentage of Participants Retained in the Study at Post Treatment
Description: Retained patients will be defined as those providing patient reported outcomes scores (e.g., pain, anxiety) at post-treatment. Separate retention rates (# retained / # enrolled) will be assessed overall and by site.
Time Frame: At post treatment (45-60 minutes)
Population: Participants who enrolled
Measure: Number; unit: percentage of patients retained at post
Groups:
- Total Enrolled: Total Enrolled across all 3 sites
- University Hospitals/Case Western: Enrolled at University Hospitals/Case Western
- VUMC: Enrolled at VUMC
- UCSD: Enrolled at UCSD
Arm/Group | Total Enrolled | University Hospitals/Case Western | VUMC | UCSD
Number analyzed (Participants) | 165 | 61 | 49 | 55
percentage of patients retained at post | 91.5 | 98.4 | 95.5 | 80

3. Secondary Outcome: Percentage of Patients Retained at 1-week Follow up
Description: Retained patients will be defined as those providing patient reported outcomes scores at 1 week. Separate retention rates (# retained / # enrolled) will be assessed overall and by site.
Time Frame: One-week after the participant was discharged from the ED
Population: Participants who enrolled
Measure: Number; unit: percentage of patients retained at 1-wk
Groups:
- Total Enrolled: Enrolled across all 3 sites
Arm/Group | Total Enrolled | University Hospitals/Case Western | VUMC | UCSD
Number analyzed (Participants) | 165 | 61 | 49 | 55
percentage of patients retained at 1-wk | 77.6 | 82.0 | 81.6 | 69.1

4. Secondary Outcome: Patient Satisfaction Question 1 at Post-treatment
Description: Question 1: "How satisfied are you with how your pain was managed during your ED visit" on the 5-point Likert scale (1-Very Satisfied; 2-Satisfied; 3-Neither Satisfied nor Dissatisfied; 4-Dissatisfied; 5-Strongly Dissatisfied).
Time Frame: At post-treatment (45-60 minutes after baseline)
Population: Participants who has Post-treatment scores and answered satisfaction question 1 at post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Total Satisfaction: Total Satisfaction across all 3 sites
- Acupuncture: Satisfaction for those randomized to acupuncture in the ED and who answered the question
- Usual Care: Satisfaction for those randomized to the Usual Care arm and who answered the question
Arm/Group | Total Satisfaction | Acupuncture | Usual Care
Number analyzed (Participants) | 140 | 69 | 71
units on a scale | 3.91 (1.23) | 4.36 (1.06) | 3.46 (1.23)

5. Secondary Outcome: Patient Satisfaction Question 2 at Post-treatment
Description: "Overall how satisfied are you with your treatment during your ED visit?" on the 5-point Likert scale (1-Very Satisfied; 2-Satisfied; 3-Neither Satisfied nor Dissatisfied; 4-Dissatisfied; 5-Strongly Dissatisfied).
Time Frame: At post-treatment (45-60 minutes after baseline)
Population: Participants who has Post-treatment scores and answered satisfaction question 2 at post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Total Satisfaction: Satisfaction across all sites
- Acupuncture: Satisfaction for those randomized to the Acupuncture Arm
- Usual Care: Satisfaction for those randomized to the Usual Care Arm
Arm/Group | Total Satisfaction | Acupuncture | Usual Care
Number analyzed (Participants) | 139 | 68 | 71
units on a scale | 4.13 (1.12) | 4.57 (0.78) | 3.70 (1.22)

6. Secondary Outcome: Patient Satisfaction Question 1 at 1-Week
Description: "How satisfied are you with how your pain was managed during your ED visit" on the 5-point Likert scale (1-Very Satisfied; 2-Satisfied; 3-Neither Satisfied nor Dissatisfied; 4-Dissatisfied; 5-Strongly Dissatisfied).
Time Frame: One week after participant was discharged from the ED
Population: Participants who has Post-treatment scores and answered satisfaction question 1 at 1-week FU
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Total Satisfaction: Satisfaction for all participants
Arm/Group | Total Satisfaction | Acupuncture | Usual Care
Number analyzed (Participants) | 133 | 69 | 64
units on a scale | 3.95 (1.27) | 4.16 (1.21) | 3.73 (1.30)

7. Secondary Outcome: Patient Satisfaction Question 2 at 1 Week
Description: as for outcome 5
Time Frame: One week after participant was discharged from the ED
Population: Participants who has Post-treatment scores and answered satisfaction question 2 at 1-week FU
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Total Satisfaction: Satisfaction across sites
Arm/Group | Total Satisfaction | Acupuncture | Usual Care
Number analyzed (Participants) | 134 | 70 | 64
units on a scale | 3.98 (1.23) | 4.19 (1.16) | 3.75 (1.27)

8. Secondary Outcome: Provider Satisfaction Question1
Description: "Do you view acupuncture in general as an appropriate intervention for the ED setting?" on a 5 point scale (0: Very inappropriate; 1: Inappropriate; 2: Neutral; 4: Appropriate; 4: Very appropriate). Higher scores are better.
Time Frame: After enrollment at the provider's site completed (~6 months after first enrollee).
Population: Providers who responded to the survey after their site completed enrollment.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Appropriateness: Average score of providers' perception of appropriateness of acupuncture in the ED
Arm/Group | Appropriateness
Number analyzed (Participants) | 125
score on a scale | 2.19 (1.07)

9. Secondary Outcome: Provider Satisfaction Question 2
Description: "Do you view acupuncture in general as helpful in managing patient pain in the ED?" on a 5 point scale (0: Not at all helpful; 1: Somewhat Unhelpful; 2: Neutral; 3: Somewhat Helpful; 4: Very Helpful). Higher scores are better.
Time Frame: After enrollment at the provider's site completed (~6 months after first enrollee).
Population: Providers who responded to the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Helpful: Average score of providers' perception of helpfulness of acupuncture in the ED
Arm/Group | Helpful
Number analyzed (Participants) | 124
score on a scale | 2.50 (1.11)

10. Secondary Outcome: Provider Satisfaction Question 3
Description: "How satisfied are you with the way that the acupuncture intervention was implemented in your setting" on the 5-point Likert scale (4-Very Satisfied; 3-Satisfied; 2-Neither Satisfied nor Dissatisfied; 1-Dissatisfied; 0-Very Dissatisfied). Higher scores are better
Time Frame: After enrollment at the provider's site completed (~6 months after first enrollee).
Population: Providers who responded to the survey and were exposed to ACUITY
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Satisfied: Of those ED providers who were exposed to ACUITY, how satisfied were they with acupuncture as delivered in the study?
Arm/Group | Satisfied
Number analyzed (Participants) | 32
score on a scale | 3.03 (0.90)

11. Secondary Outcome: Provider Satisfaction Que4
Description: "Did the ACUITY project impose a burden on ED staff in your setting?" on the 4-point Likert scale (0-Not at all a burden; 1-Somewhat of a burden; 2-Moderate burden 3-Extreme burden). Lower scores are better
Time Frame: After enrollment at the provider's site completed (~6 months after first enrollee).
Population: Providers who responded to the survey and were exposed to ACUITY
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Burden: Of those ED providers who were exposed to ACUITY, what was their perception of how much burden did the study impose in your setting?
Arm/Group | Burden
Number analyzed (Participants) | 32
score on a scale | 0.38 (0.66)

ADVERSE EVENTS:
Time Frame: Any adverse event from baseline to 4 weeks for the Acupuncture and Usual Care Arms, approximately 6 months for the ED Staff/Providers Arm
Arm/Group | Acupuncture | Usual Care | ED Staff/Providers
All-Cause Mortality (participants affected / at risk) | 1/83 | 0/82 | 0/125
Serious Adverse Events (participants affected / at risk) | 1/83 | 1/82 | 0/125
Other Adverse Events (participants affected / at risk) | 0/83 | 0/82 | 0/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acupuncture (N=83) | Usual Care (N=82) | ED Staff/Providers (N=125)
Death (Vascular disorders) | 1 (1) | 0 (0) | NA — Death due to retroperitoneal hemorrhage (preliminary cause of death) and cirrhosis (secondary) at Site 2 about 7 days after their ED discharge and subsequent inpatient admission . It was unanticipated, fatal and not study related
Hospitalization for Suspected Stroke (Vascular disorders) | 0 (0) | 1 (1) | NA — Hospitalization included diagnosis of new cerebral mass lesion concerning for metastasis and likely culprit of the patients symptoms. Patient also diagnosed with Left low extremity DVT. It was unexpected, severe and not study related

LIMITATIONS AND CAVEATS:
It should be noted that recruitment was conducted during the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-12-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT04880733/Prot_SAP_ICF_003.pdf